CLINICAL TRIAL: NCT04979312
Title: Predictive Role of Non-Invasive Glucose Assessment During Pregnancy: A Pilot Study
Brief Title: Glucose and Blood Pressure During Pregnancy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting device from Sponsor
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 21-000284
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gestational Diabetes; Pre-Eclampsia; Blood Pressure
MeSH Terms: conditions — Diabetes, Gestational; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LabClasp+Standard of care (Experimental)
  Interventions: Device: LabClasp
- Standard of care (No Intervention)

INTERVENTIONS:
Device: LabClasp — Subjects will complete up to 10 measurements per day with potentially more before and during their OGTT using the LabClasp
  Arms: LabClasp+Standard of care

SUMMARY:
The purpose of this research is to examine the beneficial effects of regular, non-invasive, glucose (sugar) assessment on glucose (sugar) and blood pressure regulation during pregnancy to help in predicting gestational diabetes and preeclampsia.

DETAILED DESCRIPTION:
This is an open-label pilot trial for the LabClasp combined with standard clinical care compared to standard clinical on [glucose] and blood pressure during pregnancy. Potential study participants will be pre-screened using questionnaires and review of their clinical records. Once the consent has been obtained, participants will undergo screening to confirm eligibility. Subjects who meet all criteria will be randomized to either LC+SC or SC cohorts for 24-39wks depending upon their gestational duration at enrollment. Study measures including anthropometrics, surveys/questionnaires, 24hr ABPM, accelerometry, and an oral glucose tolerance test (OGTT). Furthermore, the investigators will obtain repeated (annual) subject information including vitals, labs, medications, and development of cardiometabolic disorders for up to 10yrs in follow-up by reviewing Mayo Clinic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-45 years (inclusive)
* Body mass index (BMI) ≤40kg/m2
* >1 risk factor for GDM
* <16wks gestation
* Gender: only females will be recruited into this study
* Ability to provide written informed consent

Exclusion Criteria:

* Presence of chronic kidney disease (creatinine >2.5mg/dL) and/or active cancer
* Smoking
* Multiple pregnancies
* Congenital abnormalities
* Use of chronic medications which influence blood [glucose] or [insulin]
* Subsequent diagnosis of GDM or preeclampsia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant females will be recruited into this study
Enrollment: 100 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 30
  Blood Glucose will be measured in Mmol/L
Systolic Blood Pressure | Baseline
  Systolic Blood Pressure will be measured in mmHg
Diastolic Blood Pressure | Baseline
  Diastolic Blood Pressure will be measured in mmHg

SECONDARY OUTCOMES:
Pittsburgh sleep study quality index | Baseline
  The Pittsburgh Sleep Quality Index measures the severity of sleep disturbances. Possible scores range from 0 to 21 with higher scores indicating a worse outcome/more severe symptoms of sleep disturbance.

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No